CLINICAL TRIAL: NCT06490081
Title: To Evaluate the Protective Effect of Trilaciclib on Myelosuppression in Patients With Limited-stage Small Cell Lung Cancer Associated With Concurrent Chemoradiotherapy and Discuss the Effect of Gut Microbiota Changes on Myelosuppression
Brief Title: Trilaciclib Prevents Myelosuppression With Chemoradiotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4382
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-07

CONDITIONS: Myelosuppression
MeSH Terms: interventions — trilaciclib; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trilaciclib combined with concurrent chemoradiotherapy (Experimental): Trilaciclib is used simultaneously before the first cycle of chemotherapy during radiotherapy for limited-stage small cell lung cancer
  Interventions: Drug: Trilaciclib

INTERVENTIONS:
Drug: Trilaciclib — During concurrent chemoradiotherapy in limited-stage small cell lung cancer, Trilaciclib is administered prophylactically before the first cycle of chemotherapy
  Other Names: Trilaciclib combined with concurrent chemoradiotherapy

SUMMARY:
To evaluate the protective effect of Trilaciclib on myelosuppression in patients with limited-stage small cell lung cancer associated with concurrent chemoradiotherapy and discuss the effect of gut microbiota changes on myelosuppression

DETAILED DESCRIPTION:
The occurrence of myelosuppression following chemotherapy, including severe neutropenia and hematological toxicity (Grade 3/4), as well as its association with dynamic changes in the gut microbiota, was investigated in conjunction with prophylactic administration of the CDK4/6 inhibitor Trilaciclib prior to the initiation of chemotherapy during radiotherapy for limited stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The histopathology is limited-stage small cell lung cancer.
2. ECOG score 0-2.
3. Good organ function (no blood transfusions, no hematopoietic stimulating factors, no transfusions of albumin or blood products within 14 days prior to the examination).
4. It is suitable for patients treated with Trilaciclib combined with etoposide plus cisplatin or carboplatin.
5. Understand and can sign informed consent

Exclusion Criteria:

1. Brain metastases with clinical symptoms require local radiotherapy or hormone therapy.
2. Active infections require systemic treatment.
3. Subjects with active, known or suspected autoimmune disease or history of autoimmune disease.
4. Combined with other tumors.
5. The current or previous presence of a clinically significant and medically unstable condition, which in the investigator's professional judgment may compromise subject safety, interfere with study evaluation or endpoint assessment, or otherwise impact the reliability of study results.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of severe neutropenia | 14 days
  Grade 3/4 decline in neutropenia after the first cycle of chemotherapy during radiotherapy
Duration of severe neutropenia | 5 days
  Duration of severe neutropenia after the first cycle of chemotherapy during radiotherapy (ANC<1.0×10^9/L for more than 5 days)
Occurrence of hematological toxicity | 5 days
  Grade 3/4 decline in neutrophils, platelets, and red blood cells

CONTACTS AND LOCATIONS:
Overall Officials: Lei Deng, PhD, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China